CLINICAL TRIAL: NCT02815046
Title: Prospective, Non-randomized, Single-center Observational Study of Outcome Measures of Patients Suffering From Mixed Urinary Incontinence Before and After Surgical Procedure With Botulinum Toxin and Polyacrylamide Hydrogel (PAHG)
Brief Title: Mixed Urinary Incontinence Symptoms Before and After Treatment With Botox and Bulkamid
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Volker Viereck (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Volker Viereck, Professor, MD, Cantonal Hospital, Frauenfeld
Organization: Cantonal Hospital, Frauenfeld (Other)
Other Study IDs: Botox-Bulkamid study
Record Dates: First submitted 2016-06-08; First posted 2016-06-28 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Mixed Incontinence, Urge and Stress
Keywords: urgency urinary incontinence; stress urinary incontinence; Botulinum toxin A; Bulkamid
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Botulinum toxin type A — Intravesical injections of Botulinum toxin A (Botox) into the bladder wall.
  Other Names: Botox
Device: Polyacrylamide hydrogel — Midurethral injections of the bulking Agent Bulkamid into the submucosal tissues of the urethra.
  Other Names: Bulkamid

SUMMARY:
This study compares mixed urinary incontinence symptoms before and after a combined treatment with Botox and Bulkamid. Eligible for the study are adult females with a mixed urinary incontinence, having both urgency urinary symptoms and stress urinary symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥ 18 years.
2. Clinically diagnosed therapy-refractory mixed urinary incontinence (MUI) based on cough test, urodynamic evaluation, 3-day micturition diary, incontinence-questionnaire with visual analog scales for SUI and UUI.
3. All criteria for the indication to treat patient with Botox are met.
4. All criteria for the indication to treat patient with Bulkamid are met.
5. Participant has given informed consent

Exclusion Criteria:

1. All contraindications for Bulkamid or Botox
2. Previous treatment with Botulinum toxin (within last 3 months)
3. Previous treatment with Bulkamid or other bulking agent (within last 3 months)
4. Participant is pregnant or lactating
5. Current urinary tract infection (in which case this has to be treated first before patient might be included)
6. Residual urine of > 100 ml

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mixed urinary incontinence (MUI) eligible for an intervention with Botox and Bulkamid.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-08; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Cure rates for stress urinary incontinence (SUI) | 6 months
  Number of participants with negative cough stress test and 90 % improved SUI-visual analog scale.
Change from baseline in number of micturitions per day | Baseline, 6 months

SECONDARY OUTCOMES:
Frequency of complications | intra-operative and post-operative follow-up up to 12 months
Frequency of cough stress test levels | Baseline, 6 months, 12 months
  3 Levels: negative, only a few drops of urine, severe loss of urine
SUI-visual analog scale | Baseline, 6 months, 12 months
  Scale from 0-10: 0-no suffering - 10-severe suffering
UUI-visual analog scale | Baseline, 6 months, 12 months
  Scale from 0-10: 0-no suffering - 10-severe suffering
Change from baseline in number of micturitions per day | Baseline, 6 months, 12 months
Change from baseline in number of urgency episodes per day | Baseline, 6 months, 12 months
Change from baseline in number of urgency urinary incontinence episodes per 3 days | Baseline, 6 months, 12 months
Change from baseline in urine volume per micturition | Baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Volker Viereck, MD, Principal Investigator — Cantonal Hospital, Frauenfeld
Locations (1):
- Cantonal Hospital Frauenfeld, Frauenfeld, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Publication in peer-reviewed journal